CLINICAL TRIAL: NCT07360054
Title: The Effect of Virtual Reality on Pain, Anxiety, and Vital Signs During Femoral Sheath Removal After Coronary Angiography: A Randomized Controlled Trial
Brief Title: Effect of Virtual Reality on Pain, Anxiety, and Vital Signs During Femoral Catheter Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Emine Korkmaz, Principal Investigator, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VR-FEM-SHEATH-01
Record Dates: First submitted 2026-01-03; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pain; Anxiety; Hemodynamic Response; Coronary Artery Disease
Keywords: Virtual Reality, Pain Management, Anxiety, Femoral Catheter Removal
MeSH Terms: conditions — Pain; Anxiety Disorders; Coronary Artery Disease; Agnosia

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the virtual reality intervention group or the control group receiving routine care, and both groups were followed in parallel throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Participants received a virtual reality application during femoral catheter removal in addition to routine clinical care.
  Interventions: Other: Virtual Reality
- Control Group (No Intervention): Participants received routine clinical care during femoral catheter removal without any additional intervention.

INTERVENTIONS:
Other: Virtual Reality — A virtual reality application providing immersive audiovisual content was used during femoral catheter removal to reduce pain and anxiety.
  Arms: Virtual Reality Group

SUMMARY:
Femoral catheter removal after coronary angiography is a common clinical procedure that may cause pain, anxiety, and changes in vital signs in patients. Non-pharmacological interventions are increasingly used to improve patient comfort and safety during invasive procedures.

The purpose of this randomized controlled study is to evaluate the effect of a virtual reality (VR) application on pain, anxiety, and vital signs during femoral catheter removal in patients undergoing coronary angiography. Participants were randomly assigned to either a virtual reality group or a control group receiving routine care. Patients in the intervention group experienced a virtual reality application during femoral catheter removal, while the control group received standard clinical care.

Pain intensity, anxiety levels, and vital signs were assessed before, during, and after the procedure. The findings of this study are expected to contribute to evidence-based nursing practice by supporting the use of virtual reality as a safe and effective non-pharmacological method to reduce discomfort during femoral catheter removal.

DETAILED DESCRIPTION:
Coronary angiography is a widely used diagnostic procedure in cardiology, and femoral arterial access remains common in many clinical settings. Removal of the femoral catheter following the procedure is frequently associated with pain, anxiety, and physiological responses such as changes in blood pressure and heart rate. These symptoms may negatively affect patient comfort and overall procedural experience.

Virtual reality (VR) is a non-pharmacological intervention that provides immersive audiovisual stimulation and has been shown to reduce pain and anxiety by diverting attention and promoting relaxation. However, evidence regarding its effectiveness during femoral catheter removal after coronary angiography remains limited.

This single-center, randomized controlled trial was conducted to determine the effect of virtual reality on pain intensity, anxiety levels, and vital signs during femoral catheter removal in patients undergoing coronary angiography. Eligible patients were randomly assigned to either the virtual reality intervention group or the control group. Patients in the intervention group received a virtual reality application during femoral catheter removal, while patients in the control group received routine clinical care.

Data were collected using a patient information form, a visual analog scale for pain assessment, a standardized anxiety assessment tool, and vital signs monitoring. Measurements were obtained before, during, and after femoral catheter removal. The results of this study aim to provide evidence supporting the integration of virtual reality into nursing care practices to enhance patient comfort and improve the quality of care during invasive cardiovascular procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Ability to speak and understand Turkish
* Undergoing elective coronary angiography with femoral arterial access
* Planned femoral sheath removal
* Hemodynamically stable vital signs
* No psychiatric, cognitive, visual, or hearing impairment
* No administration of analgesics for any reason prior to sheath removal

Exclusion Criteria:

* Use of analgesics for chronic pain prior to the procedure
* Impaired orientation to time or place
* Use of anxiolytic and/or sedative medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity measured by Visual Analog Scale (VAS) | Before femoral sheath removal (baseline), during femoral sheath removal (procedural period), and immediately after sheath removal
  Pain intensity will be assessed using the Visual Analog Scale (VAS), scored from 0 (no pain) to 10 (worst pain). Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
Anxiety level measured by State Anxiety Inventory (STAI-S) | Before sheath removal (baseline) and immediately after sheath removal
  Anxiety will be measured using the State-Trait Anxiety Inventory - State Form (STAI-S), assessing state (situational) anxiety only.
  The scale consists of 20 items, with scores ranging from 20 (low anxiety) to 80 (high anxiety). Higher scores indicate greater anxiety.
Heart rate measured in beats per minute (bpm) | Before sheath removal (baseline), during femoral sheath removal (procedural period), and immediately after sheath removal
  Heart rate will be measured using standard clinical monitoring equipment and reported in beats per minute (bpm).
Systolic blood pressure measured in mmHg | Before sheath removal (baseline), during femoral sheath removal (procedural period), and immediately after sheath removal
  Systolic blood pressure will be measured using non-invasive monitoring and reported in millimeters of mercury (mmHg).
Diastolic blood pressure measured in mmHg | Before sheath removal (baseline), during femoral sheath removal (procedural period), and immediately after sheath removal
  Diastolic blood pressure will be measured using non-invasive monitoring and reported in millimeters of mercury (mmHg).
Respiratory rate measured in breaths per minute | Before sheath removal (baseline), during femoral sheath removal (procedural period), and immediately after sheath removal
  Respiratory rate will be measured via standard clinical observation and reported as breaths per minute.
Oxygen saturation measured by pulse oximetry (SpO₂ %) | Before sheath removal (baseline), during femoral sheath removal (procedural period), and immediately after sheath removal
  Peripheral oxygen saturation (SpO₂) will be measured using pulse oximetry and reported as percentage (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical restrictions and to protect participant confidentiality. The data are used solely for the purposes of this study.